CLINICAL TRIAL: NCT04880551
Title: Ventilation Imbalances in Mild to Moderate Chronic Obstructive Pulmonary Disease
Acronym: VAPOR
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Oregon Health and Science University (Other)
Collaborators: 4DMedical (Industry)
Responsible Party: Principal Investigator, Akram Khan, Principal Investigator, Oregon Health and Science University
Other Study IDs: IRB00022285
Record Dates: First submitted 2021-04-12; First posted 2021-05-10 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: COPD; Dyspnea; Respiratory Disease; Lung Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Respiration Disorders; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- COPD patients with a recent Spirometry: Patients that have a diagnosis of COPD and have completed a recent Pulmonary Function Test - Spirometry.
  Interventions: Radiation: Fluoroscopy

INTERVENTIONS:
Radiation: Fluoroscopy — In this study the patient will be exposed to radiation during the fluoroscopy for lungs. There is a small chance of alopecia. There is a rare chance that the patients skin may turn red or be damaged.
  Other Names: 4DXV Lung Ventilation Analysis Software (LVAS)

SUMMARY:
The Investigators plan a single center study to get preliminary data to answer a number of fundamental questions directly related to management of COPD. The research will determine whether ventilation heterogeneity and distribution of ventilation inform, determine, assist or drive the: 1) status or clinical course in patients with COPD, 2) understanding of factors associated with activities of daily living and quality of life in patients , 3) risk of exacerbation or hospitalization in those with COPD, and 4) predictors of therapeutic pathway or treatment regime.

DETAILED DESCRIPTION:
The Investigators plan a single center study to get preliminary data to answer a number of fundamental questions directly related to management of COPD. The research will determine whether ventilation heterogeneity and distribution of ventilation inform, determine, assist or drive the: 1) status or clinical course in patients with COPD, 2) understanding of factors associated with activities of daily living and quality of life in patients , 3) risk of exacerbation or hospitalization in those with COPD, and 4) predictors of therapeutic pathway or treatment regime.

Specific Aims

Aim 1: Determine if XV Lung Ventilation Analysis Software yields valid and clinically useful quantification of ventilation in COPD subjects.

The goal of aim 1 is to develop the practical and technical components to deploy XF functional lung imaging within the institution in collaboration with, pulmonary and radiology, infrastructure from information technology and administration. After initial testing, LVAS will be deployed in the institution for the study and validated against data from 4DMedical.

Aim 2: Determine if XV Lung Ventilation Analysis Software provides enhanced clinical assessment of lung function as compared to standard spirometry, SGRQ, COPD assessment test (CAT), Borg dyspnea score, mMRC questionnaire, 6MWT, and recent-CT.

In aim 2, the Investigators will take patients presenting to our outpatient clinics or recently discharged from the hospital with presence of COPD in spirometry and approach them for consenting for the study. After informed consent Investigators will collect baseline demographic data, study questionnaires and assess functional capacity using 6MWT and perform a noncontrast CT chest if not performed previously and perform fluoroscopy to get data for 4DXV lung imaging. Patients will continue with their usual pharmacological therapies and exercise program. These data points will be repeated between 4-8 weeks and 10-14 weeks to get very short-term (4-8 weeks) and short-term (10-14 weeks) changes in clinical assessment, spirometry and 4DXV lung imaging.

Aim 3: Determine the sample size for effect for future studies in COPD patients.

In aim 3, investigators will analyze data generated in aim 2 to determine if there are very short and short-term changes in spatial distribution of lung ventilation with changes in patient's clinical condition as determined by clinical assessment and spirometry to determine if the 4DXV technology can be used to study and understand progression of COPD in patients with mild to moderate disease. Data generated with the used to analyze the sample size necessary to perform a multicenter study incorporating the use of 4DXV technology in the management of patients with mild-moderate COPD and to determine what data points from the 4DXV technology can be used in clinical trials of COPD.

Each aim of the proposal will generate several products for clinical and research audiences to better understand and develop the use of 4DXV technology. The Investigators plan to develop two products using this results of the study:

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 - 85 years at Visit 1 and willing to give informed consent to participate, signed or electronic.
2. A female is eligible to enter and participate in the study if she is of:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal)
   2. Childbearing potential has a negative serum pregnancy test at Visit 1, and agrees to an acceptable method of contraception considered appropriate by patient's primary care provider.
3. COPD Diagnosis: Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) [Celli, 2004]: Progressive airflow limitation associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking.
4. Tobacco Use: Current or former smokers with a history of at least 10 pack-years of cigarette smoking. [Number of pack-years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years represent 10 pack-years)].
5. COPD Severity: Subjects with an established clinical history of COPD and severity defined as: FEV1/FVC ratio must be <0.70 and FEV1 between 40-80% of predicted normal value calculated using NHANES III reference equations.
6. Clinical data reviewed by the investigator does not suggest any harm to the patient from study enrollment.
7. Chest x-ray or computed tomography (CT) scan of the chest/lungs if available do not have clinically significant abnormalities not believed to be due to the presence of COPD
8. Compliance: Subjects must be willing to remain at the study center as required per protocol to complete all visit assessments.

Exclusion Criteria:

1. Women who are pregnant or lactating or are planning to become pregnant during the course of the study, or women of childbearing potential who are not using an acceptable method of contraception.
2. Respiratory:

   1. Asthma: Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
   2. Alpha-1 Antitrypsin Deficiency: Subjects who have alpha-1 antitrypsin deficiency as the cause of COPD.
   3. Other Respiratory Disorders: Subjects who have other active pulmonary disease such as active tuberculosis, lung cancer, significant bronchiectasis (high resolution CT evidence of bronchiectasis that causes repeated acute exacerbations), sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or uncontrolled sleep apnea (i.e., in the opinion of the Investigator severity of the disorder would impact the conduct of the study). Note: Allergic rhinitis is not exclusionary.
   4. Lung Volume Reduction: Subjects who have undergone lung volume reduction surgery, lobectomy or bronchoscopic lung volume reduction (endobronchial blockers, airway bypass, endobronchial valves, thermal vapor ablation, biological sealants, and airway implants) within 6 months of Visit 1.
   5. Hospitalization or acute COPD worsening: Subjects who have been hospitalized due to poorly controlled COPD within 2 weeks prior to Visit 1 (Screening)
   6. Chest x-ray (frontal and lateral) with suspicion of pneumonia or other condition/abnormality that will require additional investigation/treatment or put the subject at risk because of participation in the study.
3. Spirometry Performance:

   1. Acceptability: Subjects who cannot perform acceptable spirometry (i.e., meet ATS/ERS acceptability criteria)
   2. Repeatability: Subjects who cannot perform technically acceptable spirometry with at least 3 acceptable flow-volume curves with 2 or more meeting ATS repeatability criteria for FEV1 during at least 1 of the pre-bronchodilator assessments
   3. Subjects who are medically unable to withhold their short-acting bronchodilators for the six hour period prior to spirometry testing.
4. Oxygen / non-invasive positive pressure ventilation device: Subjects receiving long-term-oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 15 hours a day or using non-invasive positive pressure ventilation device. Note: Subjects using continuous positive airway pressure or bi-level positive airway pressure for Sleep Apnea Syndrome are allowed in the study if not used for ventilatory support.
5. Cardiac disease:

   1. Subjects who have unstable ischemic heart disease, left ventricular failure, or documented myocardial infarction within 6 months of enrollment.
   2. Subjects with a recent history of acute coronary syndrome, or who have undergone percutaneous coronary intervention or coronary artery bypass graft within the past 3 months are to be excluded.
   3. Subjects with congestive heart failure (CHF NYHA Class III/IV).
   4. Clinically significant abnormal ECG with conduction abnormality or arrhythmia considered significant by principal investigator.
6. Investigational drugs or devices: treatment with investigational study drug or device in another clinical study within four weeks of study enrollment.

Ages: 30 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We plan to enroll patients presenting to OHSU hospital or clinics with clinical diagnoses of COPD and a recent spirometry.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-04-25 (Estimated); Study Completion 2024-04-25 (Estimated)

PRIMARY OUTCOMES:
Quantification of imaging data | 18 months
  Determine the XV Lung Ventilation Analysis Software quantification of ventilation defect percentage and ventilation heterogeneity in COPD.
  Data will be quantified by the number of participants yielding significant ventilation defect percentages and ventilation heterogeneity in patients with COPD. Data acquired will be used to assess COPD severity using the COPD Severity Score.
Clinical Assessment of Lung Function | 18 Months
  Determine if XV Lung Ventilation Analysis Software provides enhanced clinical assessment of lung function as compared to standard spirometry, 6MWT, SGRQ and recent-CT.
Clinical assessment and correlation with imaging | 18 months
  Determine if the ventilation defect percentage and ventilation heterogeneity are associated with the change in COPD assessment test after onset of therapy. Measurements of ventilation defect percentage and ventilation heterogeneity will be compared to changes in COPD assessments during the study.
  COPD Assessments Test will be used to assess changes from Baseline measurements and 12 week assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: OHSU Pulmonary Critical Care Medicine — http://www.ohsu.edu/pccm/